CLINICAL TRIAL: NCT06695663
Title: Referral Training and eGen Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: cont
Record Dates: First submitted 2024-10-31; First posted 2024-11-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Behavioral Problem; Behavioral Problem of Child
MeSH Terms: conditions — Problem Behavior | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Primary care clinicians group 1 (Experimental): PCCs with pediatric patients randomized to experimental group
  Interventions: Behavioral: Referral and communication skills learning
- Primary care clinicians group 2 (Active Comparator): PCCs with pediatric patients randomized to control group
  Interventions: Behavioral: Written guide to the referral process
- Parent group 1 (Experimental): assigned to receive eGen
  Interventions: Behavioral: Empowered Generations (eGen): parent training
- Parents group 2 (Active Comparator): assigned to receive one-session control
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: Referral and communication skills learning — assigned to receive a brief, live, experiential training on the referral process and communication strategies.
  Arms: Primary care clinicians group 1
Behavioral: Written guide to the referral process — assigned to receive only written information about the referral process
  Arms: Primary care clinicians group 2
Behavioral: Empowered Generations (eGen): parent training — eGen is a six-session parent training program provided by therapists via video chat online to parents with a child between the ages of 3-8 years.
  Arms: Parent group 1
Behavioral: control — The control condition consists of a single scripted session, in which therapists guide the parent to the following resources: (a) a book, Raising Cooperative Kids, by GenPMTO co-developer Marion Forgatch; (b) vetted parenting advice websites; (c) information about Early Childhood and Family Education classes, which are provided for free in Minnesota through public schools; and (d) a list of culturally tailored parenting advice websites.
  Arms: Parents group 2

SUMMARY:
Child and adolescent behavioral health problems are related to the leading causes of youth morbidity and mortality. Parent-focused interventions effectively prevent behavioral health problems such as depression and conduct disorders and can provide a downstream economic benefit to society by reducing criminal activity, education costs, and health care use.

Unfortunately, parenting programs are not widely available, accessible, nor well-attended.

Pediatric primary care is a non-stigmatizing setting with nearly universal reach and, therefore, an ideal contact point to increase access. However, primary care clinicians (PCCs) often have insufficient training in behavioral health topics and typical referral practices are inadequate.

There are also logistical barriers to attending in-person parenting programs, like the need for childcare and a large time-commitment. There is a need to develop effective referral practices in conjunction with increasing the accessibility of parenting programs. The study long-term goal is to prevent significant behavioral health problems through widespread access to effective and accessible parenting programs through primary care referrals.

In this study there are two trials: First is the primary care clinicians "PCC" trial, testing the effectiveness of referral training (aim 1). Second is the parents "eGen" trial provided by therapists, testing the effectiveness of eGen parenting intervention (aim 2).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for parent in the randomized controlled trial include being a parent or caregiver of a child ages 3 to 8 and having a referral to a participating therapist from a primary care provider.
* The only inclusion criteria is that participants be a PCC who sees children between the ages of 3- 8 years old. PCCs must also have approval from their clinic to participate. Vulnerable populations will not be targeted from inclusion but may be included if they meet the previously stated inclusion criteria.

Exclusion Criteria:

* Parents would be excluded if there is a reasonable belief that participating could increase danger to a child or if they are psychologically unable to engage in the intervention activities.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Child behavior problems | 10 weeks
  Child externalizing and internalizing will be measured using the Behavioral Assessment System for Children - Behavioral and Emotional Screening System (BASC-3-BESS; 29 items).
Change in parenting behavior | 10 weeks
  The Alabama Parenting Questionnaire - Preschool version (APQ; 32 items) has subscales to measure positive parenting, inconsistent parenting, and punitive parenting.
Number of Completed Referrals | 4 years
  This is defined as the number of parents who agree to begin treatment with the therapist after a referral from a primary care provider.
Parent Attendance | 1 year
  Parent attendance will be reported as the percent of sessions attended.

SECONDARY OUTCOMES:
Parents mental health: depression | 10 weeks
  The patient health questionnaire will measure parent depression (PHQ-9; 9 items)
Parents mental health: anxiety | 10 weeks
  the general anxiety disorder scale (GAD-7) will assess parent anxiety symptoms
Parents mental health: absenteeism | 10 weeks
  the WHO Health and Work Performance Questionnaire - Short Form (HPQ SF, 8 items) will assess parent absenteeism.
Parenting self-efficacy | 10 weeks
  Parenting self-efficacy will be measured with the Parent Locus of Control measure (PLOC; 24 items).
Intervention Acceptability, Appropriateness, and Feasibility Measure | 1 year
  Average score on the Acceptability of intervention Measure items. These measures are on a 1-5 scale from completely disagree to completely agree. A higher score indicates higher acceptability, appropriateness, or feasibility.
Readiness to Change - Patient Preferences Subscale Score | 1 year
  Average score on the Readiness to Change Assessment, patient preferences items (Helfrich, Li; Sharp, 2009). This measure is rated on a 1-5 scale from strongly disagree to strongly agree, with a sixth option for not applicable. High scores indicates greater acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Mehus, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States